CLINICAL TRIAL: NCT07320846
Title: Investigation of the Effects of Standard Rehabilitation Program and Inspiratory Muscle Training on lncRNA HOTAIR Expression in Patients With Rheumatoid Arthritis
Brief Title: The Effect of Exercise Training on lncRNA Expression in Rheumatoid Arthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Zeynep Betül Özcan, Principal Investigator, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rheumatoid_HOTAIR; 2024-93 (Other Grant/Funding Number: Scientific Research Coordination Unit)
Record Dates: First submitted 2025-12-03; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-01

CONDITIONS: Exercise; Pulmonary Rehabilitation; Interstitial Lung Disease; Long Noncoding RNA; Inspiratory Muscle Training; Rheumatoid Arthritis
Keywords: inspiratory muscle training; long noncoding RNA; exercise; pulmonary rehabilitation; Interstitial lung disease; rheumatoid arthritis
MeSH Terms: conditions — Motor Activity; Lung Diseases, Interstitial; Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standart Pulmonary Rehabilitation Group (SGr) (Active Comparator): In the SGr program, exercises are planned to be performed under the supervision of a remote physiotherapist, 2 days a week with the telerehabilitation method and 1 day as a home- based program by the patient. The exercise program includes aerobic, resistance exercises and respiratory exercises, and patients are followed for 3 months.
  Interventions: Behavioral: Standard pulmonary rehabilitation programme
- Pulmonary Rehabilitation Group with Inspiratory Muscle Training (IGr) (Experimental): In the IGr program, exercises are planned under the supervision of a remote physiotherapist, with the telerehabilitation method 2 days a week and with a program to be done by the patient at home 1 day a week. The exercise program includes aerobics, resistance exercises, respiratory exercises and respiratory muscle strengthening training with a resistive thereshold inspiratory muscle strengthening device, and patients are followed for 3 months.
- Control Group (CGr) (Other): The KGr group will consist of women and men aged between 18-75, who have signed the informed consent form regarding the study, have a BMI <30, are non-smokers, have no known systemic disease, and have FEV1>80, and are age and gender matched to the exercise groups.
  Interventions: Other: No intervention

INTERVENTIONS:
Behavioral: Standard pulmonary rehabilitation programme — Patients are asked to perform thoracic, diaphragmatic breathing, and lower basal breathing exercises with 10 repetitions. Then, strengthening exercises are performed on the major muscle groups of the upper and lower extremities. In accordance with the resistance training program in the ATS/ERS guidelines for pulmonary rehabilitation, two to four sets of 6-12 repetitions are performed with intensities ranging from 50% to 85% of one maximum repetition, two to three times a week. During the exercises, the patient is questioned about their fatigue and dyspnea levels using the Borg scale, and breaks are given when necessary. The aerobic exercise program is performed as a 12-week, 3-day-a-week self-walking exercise. The walking program is performed in the form of walking on flat ground at 60% workload, based on the data obtained from the 6-minute walking test result (land-based walking).
  Arms: Standart Pulmonary Rehabilitation Group (SGr)
Device: Resistive threshold inspiratory muscle training — In the other arm of the study, respiratory muscle training is performed in addition to the "standard pulmonary rehabilitation program." Respiratory muscle strengthening training is performed with a resistive thereshold inspiratory muscle strengthening device. The exercise is performed at an intensity of 30% of the maximum inspiratory pressure determined by mouth pressure measurement. The exercise is performed in 7 sets, with 2 minutes of work and 1 minute break for a total of 21 minutes.
Other: No intervention — Peripheral blood samples will be taken once from the participants in the control group and no other intervention will be performed.
  Arms: Control Group (CGr)

SUMMARY:
The goal of this observational study is to examine the effects of traditional respiratory rehabilitation and respiratory muscle strengthening training added to this program at the genetic level in in patients with rheumatoid arthritis-associated interstitial lung disease. The main questions it aims to answer are:

* Does respiratory muscle strengthening exercise added to respiratory rehabilitation in patients with rheumatoid arthritis-associated interstitial lung disease have additional benefits on rehabilitation outcome measures such as exercise capacity, shortness of breath, and muscle strength?
* Does the gain obtained with respiratory muscle strengthening iin patients with rheumatoid arthritis-associated interstitial lung disease increase the quality of life of patients and have a positive effect on their psychological state?
* Does respiratory rehabilitation applied to iin patients with rheumatoid arthritis-associated interstitial lung disease have an effect on genetic changes?
* Does respiratory muscle strengthening training applied in addition to respiratory rehabilitation in patients with rheumatoid arthritis-associated interstitial lung disease have an effect on genetic changes?
* Participants will be included in two different respiratory rehabilitation programs with and without respiratory muscle training, and pre- and post- treatment rehabilitation criteria and genetic changes will be compared.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a systemic, inflammatory, and autoimmune disease characterized by inflammation of synovial tissue in the joints, which can lead to joint destruction. Although the pathogenesis of the disease is not yet fully understood, it is thought that genetic and environmental factors contribute to the pathological activation of the immune system. The presence of autoantibodies has been demonstrated in the serum of RA patients, including rheumatoid factor (RF), anti-citrullinated protein antibodies (ACPA), anti-carbamylated protein antibodies, and anti-acetylated protein antibodies. The presence of these autoantibodies provides critical insights into the pathophysiology of the disease. RA follows an inflammatory pathway characterized by the overexpression of proinflammatory cytokines. Specifically, TNF-α, IL-6, and IL-1b play significant roles in triggering joint destruction and synovial inflammation, ultimately leading to bone erosion and cartilage damage.

In addition to joint involvement, RA can also involve extra-articular organs and tissues, which may lead to significant increases in morbidity and mortality. The lungs are the primary organ affected by extra-articular involvement in RA. Pulmonary involvement in RA negatively impacts prognosis and often necessitates treatment modification. Pulmonary manifestations can present as pleural, parenchymal, or vascular involvement. Among the types of pulmonary involvement associated with RA, interstitial lung disease (ILD) is one of the most common parenchymal manifestations. However, the prevalence of ILD in RA (RA-ILD) patients varies depending on the diagnostic methods used and the populations studied. Studies have shown that ILD significantly worsens the overall prognosis of RA and often requires specific therapeutic approaches, including modifications to immunosuppressive treatments or the addition of antifibrotic therapies.

Respiratory dysfunction in RA is not solely limited to parenchymal damage. Inflammatory involvement of respiratory muscles, as well as reduced pulmonary function due to systemic inflammation, are common findings. Pulmonary function tests (PFT) in RA patients often reveal restrictive or obstructive patterns, with significant reductions in forced vital capacity (FVC) and diffusing capacity for carbon monoxide (DLCO). Moreover, seropositive RA patients, particularly those with high titers of RF or ACPA, are more likely to exhibit pulmonary abnormalities compared to seronegative patients. Factors such as age, smoking status, disease duration, and body mass index also contribute to variations in PFT outcomes.

The primary treatment goals for RA patients are remission or achieving a state of low disease activity. Disease-modifying antirheumatic drugs (DMARDs) and biological agents are employed to meet these objectives. These therapies aim to suppress systemic inflammation, reduce joint damage, and prevent extra-articular complications. In addition to pharmacological treatments, exercise training is recommended to improve patients' quality of life, enhance functional recovery, and reduce cardiovascular risks. Aerobic and resistance exercises have been shown to be both feasible and effective for RA patients, significantly improving muscle strength, joint mobility, and overall physical function without exacerbating disease activity.

Particularly in RA patients with pulmonary involvement, respiratory exercises are gaining attention for their potential to improve respiratory muscle strength and pulmonary function. Studies on respiratory training have demonstrated improvements in inspiratory and expiratory muscle strength, as well as reductions in dyspnea severity. These interventions are especially beneficial in patients with coexisting ILD, where optimizing pulmonary function can contribute to better clinical outcomes and quality of life.

LncRNA HOTAIR, a long non-coding RNA known as a repressor of the HOXD gene, has been shown to play a critical role in RA. HOTAIR facilitates inflammatory reactions by releasing inflammatory cellular contents into circulation and contributes to cartilage and bone matrix destruction through the activation of MMP-2 and MMP-9 in osteoclasts. Analyses in RA patients have demonstrated elevated HOTAIR expression levels, which have been associated with disease pathogenesis. The positive correlation between HOTAIR and TNF-α further underscores its impact on inflammation. Additionally, HOTAIR has been shown to enhance the production of MMP-9 and other matrix metalloproteinases, contributing to joint destruction.

In recent years, studies investigating the role of epigenetic modifications in the diagnosis, treatment, and progression of RA have gained increasing attention. Long non-coding RNAs (lncRNAs), which are RNA molecules longer than 200 nucleotides that do not code for proteins, are emerging as significant regulators in various biological and pathological processes. LncRNAs influence epigenetic modifications, transcription, post-transcriptional processes, and protein-RNA interactions. Some lncRNAs exhibit oncogenic properties, while others act as tumor suppressors depending on their expression profiles and biological effects in different tissues. In RA, specific lncRNAs, including HOTAIR, have been identified as key players in the inflammatory response and disease progression.

Despite the growing body of research on lncRNAs in autoimmune diseases, no studies to date have investigated the impact of exercise training on the regulation of lncRNA HOTAIR in RA-ILD patients. Given the increasing evidence linking lncRNAs to immune regulation and inflammation, understanding how exercise influences these molecules could provide novel insights into RA management. Our study aims to fill this gap by exploring the relationship between exercise training and lncRNA HOTAIR expression in RA patients, with a particular focus on the potential epigenetic mechanisms underlying these interactions. By addressing this unexplored area, we aim to contribute to the development of innovative therapeutic strategies that combine pharmacological treatments with exercise-based interventions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with RA according to the ACR/EULAR 2010 classification criteria
* Duration of diagnosis greater than 2 years
* Disease activity with a DAS28 score below 5.1
* Voluntary participation in the study
* Presence of lung involvement

Exclusion Criteria:

* Having orthopedic deformities that may affect the treatment program
* Pregnancy
* Uncontrolled diabetes or heart disease
* Participation in a rehabilitation program within the last 6 months
* Body Mass Index (BMI) > 30
* Patients with severe organ failure
* Recent acute coronary syndrome
* Presence of active infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-05-18 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2026-03-12 (Estimated)

PRIMARY OUTCOMES:
lncRNA HOTAIR expression levels | Baseline and 12 weeks
  Peripheral blood mononuclear cells (PBMCs) will be isolated from venous blood samples collected at baseline and at Week 12. Total RNA will be extracted from PBMCs and reverse-transcribed into complementary DNA (cDNA). lncRNA HOTAIR expression will be quantified using real-time quantitative polymerase chain reaction (RT-qPCR). Each sample will be analyzed in duplicate. Cycle threshold (Ct) values will be normalized to a reference housekeeping gene to calculate ΔCt values. Changes in HOTAIR expression between baseline and Week 12 will be determined using the ΔΔCt method and expressed as fold change (2-ΔΔCt).
Short Form - 36 | Baseline and 12 weeks
  In the evaluation with the short form-36, it is aimed to learn the patient's views about her own health, how she feels and how much she can perform her daily activities. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Respiratory Muscle Strength Measurement | Baseline and 12 weeks
  The patient is seated in a straight-backed chair. The patient is asked to grasp the silicone mouthpiece with his/her mouth and inhale and exhale as quickly and deeply as possible. The measurements are repeated until 3 measurement values are obtained with a maximum of 10% deviation between the measured peak value. The maximum value is taken among the measured values.
Visual Analog Scale (VAS) | Baseline and 12 weeks
  Pain level will be assessed using with Visual Analog Scale. VAS is a scale which consists of a 100-millimetre scale ranging from 0 (no pain at all) to 100 (worst imaginable pain). A higher score indicates greater pain intensity.
Exercise capacity (6-minute walk test) | Baseline and 12 weeks
  6-minute walk test is performed for exercise capacity. After resting in a chair for a sufficient period (>30 minutes), patients walk as fast as possible, without running, for 6 minutes on a straight 30-meter corridor. Before and after the test, the patient's fatigue and dyspnea are questioned using the Modified Borg Scale. Oxygen saturation and heart rate are monitored and recorded using a finger pulse oximeter before, during, and after the test.

SECONDARY OUTCOMES:
Modified Medical Research Council (mMRC) Dyspnea Scale | Baseline and 12 weeks
  mMRC is a 0-4 point category scale where patients select the value that best describes their level of dyspnea. Increases in mMRC levels, especially values of 2 and above, are considered to indicate an increased risk of mortality.
HAQ | Baseline and 12 weeks
  Health Assessment Questionnaire was used to assess general health. It consists of 20 questions in total, including 8 subsections. Subjects score between 0-3 according to their level of difficulty in activities. The total score is obtained by calculating the arithmetic mean of the sums of the highest scores in the subsections. Higher scores indicate higher functional disability and pain.
Forced Expiratory Volume in 1 Second (FEV₁) | Baseline and 12 weeks
  Change in forced expiratory volume in one second (FEV₁), measured in liters (L), assessed by spirometry using the Pony Fx spirometry device in accordance with ATS guidelines.
Forced Vital Capacity (FVC) | Baseline and 12 weeks
  Change in forced vital capacity (FVC), measured in liters (L), assessed by spirometry using the Pony Fx spirometry device in accordance with American Thoracic Society (ATS) guidelines
Quality of life level | Baseline and 12 weeks
  Saint George Respiratory Questionaire (SGRQ) score: The SGRQ ranges from 0 (no impairment of quality of life) to 100 (highest impairment of quality of life).
International Physical Activity Questionnaire-Short form (IPAQ-SF) | Baseline and 12 weeks
  It is an internationally valid questionnaire for the assessment of physical activity. The short form of the questionnaire consists of seven questions and provides information about the time spent in sitting, walking, moderate and intense activities. A score is obtained as "MET-minutes/week" by multiplying minutes, days and MET values. The numerical values obtained are classified as inactive, minimally active or very active.
Digital muscle strength measurement | Baseline and 12 weeks
  Muscle strength is assessed using an electronic hand dynamometer. The patient is asked to maintain muscle strength against the dynamometer for at least 5 seconds in each attempt, with the force measurement repeated 3 times. The best value from the 3 test results is recorded.
FEV₁/FVC Ratio | Baseline and 12 weeks
  Change in the FEV₁/FVC ratio, expressed as a percentage (%), assessed by spirometry according to ATS guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Esra PEHLİVAN, Assoc. Prof., Study Chair — Saglik Bilimleri Universitesi; Erdoğan ÇETİNKAYA, Prof. Dr., Study Director — Yedikule Chest Diseases And Thoracic Surgery Training And Research Hospital; Zeynep Betül ÖZCAN, PhD (c), Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- University of Health Sciences, Istanbul, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No